CLINICAL TRIAL: NCT05528536
Title: Investigation of the Effect of Acceptance and Commitment Therapy and Exercise in Older Adults With Chronic Pain: A Randomized Controlled Trial
Brief Title: Acceptance and Commitment Therapy and Exercise for Older Adults With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other); Aberdeen Kai-fong Welfare Association (Other); Caritas Medical Centre, Hong Kong (Other); Hong Kong Sheng Kung Hui Welfare Council Limited (Other); Hong Kong Young Women's Christian Association (Other); Neighbourhood Advice-Action Council (Other)
Responsible Party: Principal Investigator, Professor Terry Y.S. Lum, Henry G. Leong Professor in Social Work and Social Administration; Principal Investigator of the JC JoyAge project, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA200132
Record Dates: First submitted 2022-02-11; First posted 2022-09-06 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain; Older Adults; Acceptance and Commitment Therapy; Exercise; Psychosocial Intervention; Art
MeSH Terms: conditions — Chronic Pain; Motor Activity | interventions — Acceptance and Commitment Therapy; Reproductive Techniques, Assisted; Exercise; Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acceptance and Commitment Therapy (ACT) and Exercise (Experimental): This group receives eight weeks' Acceptance and Commitment Therapy (ACT) and exercise intervention.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Other: Exercise
- Art and Exercise (Sham Comparator): This group receives eight weeks' art workshops (skill-based) and exercise intervention.
  Interventions: Other: Art; Other: Exercise
- Treatment as usual (Active Comparator): This group receives treatment as usual in the local community setting.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — A two-hour ACT will focus on enhancing participant's psychological flexibility towards pain. All sessions will be delivered face-to-face within their local community centre.
  Arms: Acceptance and Commitment Therapy (ACT) and Exercise
Other: Art — To be comparable with the experimental group, the Art session will be a two-hour long session which aims to share different art techniques, without any active components. All sessions will be delivered face-to-face within their local community centre.
  Arms: Art and Exercise
Other: Exercise — An hour of low-to-moderate resistance exercise aims to increase their strength and balance. All sessions will be delivered face-to-face within their local community centre.
  Arms: Acceptance and Commitment Therapy (ACT) and Exercise; Art and Exercise
Other: Treatment as usual — treatment as usual within their community centres
  Arms: Treatment as usual

SUMMARY:
The goal of this trial is to learn if combining Acceptance and Commitment Therapy (ACT) and exercise works to reduce pain intensity, pain interference, and depressive symptoms in older adults with chronic pain and depressive symptoms.

Researchers will compare ACT + exercise intervention (ACEx) to ACT + art intervention (Art+Ex) and usual care to see if ACT + exercise intervention works to reduce pain intensity, pain interference, and depressive symptoms.

Participants will receive ACEx program, Art+Ex program, or usual care for 8 weeks and complete tests before and after the programs.

ELIGIBILITY:
Inclusion Criteria:

* age 60 years or above; and
* have depressive symptoms of mild level or above (PHQ > 5)
* have chronic pain (>3 months)
* able to give informed consent to participate

Exclusion Criteria:

* known history of autism, intellectual disability, schizophrenia-spectrum disorder, bipolar disorder, Parkinson's disease, or dementia
* (temporary exclusion criteria) imminent suicidal risk difficulty in communication
* have had stroke, fracture, cardiovascular disease, cardiovascular surgery, artery disease, surgery on vertebrae, and knee replacement in the past 6 months
* physical activity prohibited by a medical professional

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline pain intensity and interference at 8 weeks | Baseline(T0) and 8 weeks after baseline (T1)
  Brief pain inventory (BPI) is used to measure pain intensity and interference, it is a 11 items scale, using an 11-point rating, of which 0 indicates not interference and 10 as interferes completely. The higher the numbers, the greater the pain intensity and pain interference.
Change from baseline depression at 8 weeks | Baseline(T0) and 8 weeks after baseline (T1)
  The Patient Health Questionnaire (PHQ-9) is used to measure depression, it is a 9-item instrument, PHQ-9 scores of 5-9, 10-14, 15-19, 20 and above represent mild, moderate, moderately severe, and severe depression. Scores range between 0 and 27.

SECONDARY OUTCOMES:
Change from baseline anxiety at 8 weeks | Baseline(T0) and 8 weeks after baseline (T1)
  The Generalised Anxiety Disorder (GAD-2) is used to measure anxiety, it is a 2-item scale, each item is rated on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day), where higher scores indicate higher anxiety levels. Scores range between 0 and 21.
Change from baseline psychological flexibility at 8 weeks | Baseline(T0) and 8 weeks after baseline (T1)
  The Comprehensive Assessment of Acceptance and Commitment Therapy Processes (CompACT-SF) scale is used to measure psychological flexibility, it is an 8-items scale, using a 7-point rating of which 0 represents strongly disagree and 6 as strongly agree. Higher scores represent higher psychological flexibility. 3 subscales: Value Action Subscale, Openness to Experience, Behavioural Awareness, of which questions 2,3,4,7 are reverse scored.
Change from baseline pain self-efficacy at 8 weeks | Baseline(T0) and 8 weeks after baseline (T1)
  The Pain Self-Efficacy Questionnaire (PSEQ-2) is used to measure pain self-efficacy. It is a 2-items self-report, 7-point scale ranging from 0 (not at all confident) to 6 (completely confident), of which higher scores indicate stronger self-efficacy. Max score 12
Change from baseline health-related quality of life at 8 weeks | Baseline(T0) and 8 weeks after baseline (T1)
  The 12-Item Short-Form Survey (SF-12) is used to measure health-related quality of life, it is a 12 items scale, consisting of 2 subscales: Physical component score (PCS) and Mental component score (MCS). Max. score 100, higher scores indicate better physical functioning and mental health.
Change from baseline gait speed at 8 weeks | Baseline(T0) and 8 weeks after baseline (T1)
  Time up and go (TUG) is used to measure gait speed. A chair with handles is placed 3m away from an obstacle, participants are instructed to rise from the chair without touching the handles, walk to the point then return to the chair in a seated position as quickly as possible. The rating is based on the number of seconds it takes for the individual to return to the initial position where: less than 10 sec. is normal, less than 20 sec. is independent and can displace without aid, and lastly, less than 30 sec. demonstrates that that individual has difficulty walking and requires assistance with daily activity.
Change from baseline physical balance at 8 weeks | Baseline(T0) and 8 weeks after baseline (T1)
  A modified 4-Stage balanced test is used to measure physical balance, it requires the individual to stand in 4 different positions progressively for 10 seconds each. The 4 positions include: stand with feet side-by-side, place the instep of one foot next to the other foot's big toe, tandem stand, and stand with one foot. If the tandem stand cannot be held for 10 sec. indicates that the elderly is at risk of falling.
Change from baseline lower body strength at 8 weeks | Baseline(T0) and 8 weeks after baseline (T1)
  30 seconds sit to stand test is used to measure lower body strength. The participants are instructed to sit in the middle of the chair (17 inches from the ground) with hands across the chest and both feet flat on the ground. With the back straight, the participants are to rise from the chair to a standing position and then return to the sitting position for 30 seconds. The score is compared with the norm to evaluate the risk of falls.
Change from baseline upper body functioning at 8 weeks | Baseline(T0) and 8 weeks after baseline (T1)
  Grip Strength is used to measure upper body functioning. The individual is asked to sit with their back straight and arms straight on the side. The dynamometer set at the second handle will be squeezed as hard as possible alternating hands after trial. 2 trials will be taken on each hand and the sum of it will be calculated. The results will be compared to the norms to determine the participant's level of upper body functioning
Change from baseline aerobic fitness at 8 weeks | Baseline(T0) and 8 weeks after baseline (T1)
  2-min step test is used to test aerobic fitness. The individual is instructed to lift their knee to the height halfway between the iliac crest and to the patella for a total of 2 minutes. The score is the number achieved with the right knee throughout 2 minutes at the given height. The scores will then be compared to norms to determine the participant's level of aerobic fitness

OTHER OUTCOMES:
Pain intensity and interference at 3-month follow up | 20 weeks after baseline (T2)
  Brief pain inventory (BPI) is used to measure pain intensity and interference, it is a 11 items scale, using an 11-point rating, of which 0 indicates not interference and 10 as interferes completely. The higher the numbers, the greater the pain intensity and pain interference.
Depression at 3-month follow up | 20 weeks after baseline (T2)
  The Patient Health Questionnaire (PHQ-9) is used to measure depression, it is a 9-item instrument, PHQ-9 scores of 5-9, 10-14, 15-19, 20 and above represent mild, moderate, moderately severe, and severe depression. Scores range between 0 and 27.
Anxiety at 3-month follow up | 20 weeks after baseline (T2)
  The Generalised Anxiety Disorder (GAD-2) is used to measure anxiety, it is a 2-item scale, each item is rated on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day), where higher scores indicate higher anxiety levels. Scores range between 0 and 21.
Psychological flexibility at 3-month follow up | 20 weeks after baseline (T2)
  The Comprehensive Assessment of Acceptance and Commitment Therapy Processes (CompACT-SF) scale is used to measure psychological flexibility, it is an 8-items scale, using a 7-point rating of which 0 represents strongly disagree and 6 as strongly agree. Higher scores represent higher psychological flexibility. 3 subscales: Value Action Subscale, Openness to Experience, Behavioural Awareness, of which questions 2,3,4,7 are reverse scored.
Pain self-efficacy at 3-month follow up | 20 weeks after baseline (T2)
  The Pain Self-Efficacy Questionnaire (PSEQ-2) is used to measure pain self-efficacy. It is a 2-items self-report, 7-point scale ranging from 0 (not at all confident) to 6 (completely confident), of which higher scores indicate stronger self-efficacy. Max score 12
Health-related quality of life at 3-month follow up | 20 weeks after baseline (T2)
  The 12-Item Short-Form Survey (SF-12) is used to measure health-related quality of life, it is a 12 items scale, consisting of 2 subscales: Physical component score (PCS) and Mental component score (MCS). Max. score 100, higher scores indicate better physical functioning and mental health.
Gait speed at 3-month follow up | 20 weeks after baseline (T2)
  Time up and go (TUG) is used to measure gait speed. A chair with handles is placed 3m away from an obstacle, participants are instructed to rise from the chair without touching the handles, walk to the point then return to the chair in a seated position as quickly as possible. The rating is based on the number of seconds it takes for the individual to return to the initial position where: less than 10 sec. is normal, less than 20 sec. is independent and can displace without aid, and lastly, less than 30 sec. demonstrates that that individual has difficulty walking and requires assistance with daily activity.
Physical balance at 3-month follow up | 20 weeks after baseline (T2)
  A modified 4-Stage balanced test is used to measure physical balance, it requires the individual to stand in 4 different positions progressively for 10 seconds each. The 4 positions include: stand with feet side-by-side, place the instep of one foot next to the other foot's big toe, tandem stand, and stand with one foot. If the tandem stand cannot be held for 10 sec. indicates that the elderly is at risk of falling.
Lower body strength at 3-month follow up | 20 weeks after baseline (T2)
  30 seconds sit to stand test is used to measure lower body strength. The participants are instructed to sit in the middle of the chair (17 inches from the ground) with hands across the chest and both feet flat on the ground. With the back straight, the participants are to rise from the chair to a standing position and then return to the sitting position for 30 seconds. The score is compared with the norm to evaluate the risk of falls.
Upper body functioning at 3-month follow up | 20 weeks after baseline (T2)
  Grip Strength is used to measure upper body functioning. The individual is asked to sit with their back straight and arms straight on the side. The dynamometer set at the second handle will be squeezed as hard as possible alternating hands after trial. 2 trials will be taken on each hand and the sum of it will be calculated. The results will be compared to the norms to determine the participant's level of upper body functioning
Aerobic fitness at 3-month follow up | 20 weeks after baseline (T2)
  2-min step test is used to test aerobic fitness. The individual is instructed to lift their knee to the height halfway between the iliac crest and to the patella for a total of 2 minutes. The score is the number achieved with the right knee throughout 2 minutes at the given height. The scores will then be compared to norms to determine the participant's level of aerobic fitness

CONTACTS AND LOCATIONS:
Overall Officials: Terry Y.S. Lum, PhD, Principal Investigator — Department of Social Work and Social Administration, The University of Hong Kong; Gloria Wong, PhD, Principal Investigator — School of Psychology and Clinical Language Sciences, University of Reading
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT05528536/Prot_001.pdf